CLINICAL TRIAL: NCT06455397
Title: Implementing BEAM: An mHealth Tool to Prevent Mental Health Problems and Improve Developmental Outcomes in Young Children
Brief Title: Building Emotional Awareness and Mental Health (BEAM) 2024-2027
Acronym: BEAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leslie E. Roos (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Manitoba Centre for Health Policy (Unknown); George & Fay Yee Centre for Healthcare Innovation (Unknown); Children's Hospital Research Institute of Manitoba (Other); Family Dynamics, Manitoba, Canada (Unknown)
Responsible Party: Sponsor-Investigator, Leslie E. Roos, Assistant Professor, Departments of Psychology & Pediatrics, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEAM 2024-2027
Record Dates: First submitted 2024-05-29; First posted 2024-06-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Depression, Anxiety; Anger; Parenting; Stress, Psychological; Parent-Child Relations; Child Development
Keywords: Parenting; Mental health; Depression; Anxiety; Psychoeducation; App-based intervention
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress, Psychological; Psychological Well-Being | interventions — Mental Health

STUDY DESIGN:
Intervention Model Description: All study participants will complete 12 weeks of the BEAM program. This involves weekly mental health and parenting education videos, app-based social support forum, and check ins with a peer parent coach. Participants will additionally have access to systems navigation to help participants find community supports. Assessments of parent and child symptoms will occur at pre-test before BEAM begins (T1), immediately after the last week of the BEAM intervention (post-test, T2), 6-month follow-up (T3), and 12-month follow-up (T4).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The BEAM Program Group (Experimental): All study participants will complete 12 weeks of the BEAM program. Each week of BEAM includes: (a) 15-20 minutes of therapeutic mental health and parenting video content, (b) exercises to practice key skills, (c) access to the online forum to cultivate social support through interaction with other parents and peer coaches, (d) individual check ins with peer coaches (i.e., trained and supervised staff with lived experience) via Zoom for Healthcare, phone, or direct messaging, and (e) a brief in-app survey for symptom monitoring to track progress. Participants will also be invited to virtual group drop-in sessions facilitated by peer coaches and be connected with a systems navigator who can support participants in accessing other community resources (e.g., childcare programs, legal aid, housing). Co-parents will have access to all components of the BEAM program except for (d).
  Interventions: Behavioral: The Building Emotional Awareness and Mental Health (BEAM) Program

INTERVENTIONS:
Behavioral: The Building Emotional Awareness and Mental Health (BEAM) Program — The BEAM Program builds on mHealth best practices and evidence-based program design principles with the core objectives of improving maternal mental health and fostering supportive parenting. Program content draws on transdiagnostic emotion-focused mental health and third wave Cognitive Behavioural Therapy principles such as Dialectical Behavioural Therapy, Acceptance and Commitment Therapy, and the Unified Protocol.
  Program delivery will be facilitated through a mobile application. The BEAM program uses a stepped care model to address the pressing need for accessible and effective mental health interventions. Stepped care is a framework that provides mental health services in a tiered manner, ensuring that participants receive appropriate levels of support based on the severity of needs. At the heart of this model are BEAM peer coaches, who will have the most direct contact with participants. Peer coaches are trained to escalate concerns to the program clinical team as required.

SUMMARY:
Children are highly sensitive to adversity during their first five years of life, with exposure to chronic parental mental illness (MI) consistently linked to socio-emotional impairments and mental health problems in children. Children born during the COVID-19 pandemic were exposed to unprecedented level of parental distress, with parental MI reported at three times the pre-pandemic rates. This situation underscored a pressing need for scalable solutions to foster positive mental health and developmental outcomes for a generation of children. In response, the investigators developed the Building Emotional Awareness and Mental Health (BEAM) program, an innovative mobile health (mHealth) solution for parents of young children. Clinical trials to date evaluating BEAM have shown promising results, demonstrating reductions in parent depression, anxiety, and harsh parenting practices. This trial involves an effectiveness-implementation hybrid design with co-primary aims of (1) determining BEAM's effectiveness in improving child mental health and developmental outcomes, and (2) evaluating the implementation of BEAM in the community through metrics such as feasibility, acceptability, and uptake. The secondary aim of this trial is to measure BEAM's effectiveness in improving long-term biopsychosocial family outcomes using administrative data. A final exploratory aim of this trial will measure the cost-utility of delivering BEAM relative to extant health programming.

This trial will evaluate the effectiveness of implementing the BEAM intervention in the community with a sample of 400 parent participants with a child aged 24-71 months. Study participants will complete 12 weeks of psychoeducation modules in the BEAM app, with access to an online social support forum and check ins with a peer coach. Assessments of parent and child symptoms will occur at pre-test before BEAM begins (T1), immediately after the last week of the BEAM intervention (post-test, T2), 6-month follow-up (T3), and 12-month follow-up (T4).

Beginning in 2025, the trial offers participants the option to invite one parenting partner to join them in the program. A parenting partner is defined as a co-parent (e.g., the child's mother, father, or step-parent) or another primary caregiver (e.g., a grandparent, cousin, uncle, or aunt). Each participant may invite one such individual, hereafter referred to as a "co-parent." Co-parents will have access to the BEAM intervention and all its features, with the exception of peer coaching. Co-parents will be eligible to complete the same outcome measures at the same timepoints as participants. Three differences that will separate co-parents from participants are: (1) co-parents will not be asked to complete the ASQ:2-SE or ASQ-3 secondary outcome measures; (2) co-parents will not have access to peer coaching, and (3) co-parents will not be required to be experiencing moderate to severe symptoms of depression, anxiety, parenting stress, and/or anger. (Please see Eligibility > Eligibility Criteria for the less restrictive inclusion and exclusion criteria for co-parents.) Co-parents will not be counted toward the trial sample size of n=400, and will not be included in primary analyses. Instead, co-parent data will be used in sub-studies to address exploratory research questions.

The BEAM program offers a promising solution to addressing elevated parental mental health symptoms, parenting stress, and related child functioning concerns. The present implementation trial aims to extend the groundwork established by an open pilot trial and RCT of the BEAM program, in a next step of testing BEAM's readiness for nationwide scaling.

DETAILED DESCRIPTION:
The initial five years of a child's life mark a critical developmental phase and a period of high sensitivity to environmental stressors, including the impact of parental mental illness (MI) and parenting stress. Research has consistently linked parental MI with a broad range of child-related issues, including irritability, sleep disturbances, and socio-emotional developmental impairments. These adverse outcomes are often attributed to environmental factors, including parental modeling of maladaptive emotion coping strategies such as avoidance and aggression and harsh parenting practices characterized by reactive discipline and conflictual interactions. Notably, when parental MI is accompanied by additional stressors such as domestic conflict or financial strains, the long-term risks for children are exacerbated. Further, the chronicity of parental MI has critical implications for children. When stressors and parental MI are persistent, the risk of adverse developmental outcomes for children increases, putting children at heightened risk for stress and development of their own psychopathology. This highlights the critical need for interventions that address parental MI and the broader spectrum of parenting stress and its multifaceted impacts on children.

Despite the need for parents to improve their stress and mental health symptoms, the majority of parents do not access evidence-based treatments. Previous research has documented many barriers preventing parents from accessing care. These barriers include service backlogs, long waitlists, high costs of individual therapy, lack of information of where to access interventions, and overwhelming childcare demands. Additionally, although evidence-based treatments exist, most interventions do not comprehensively address the mental health of both parents and children. This gap in services is significant, given meta-analytic evidence indicating that dual-generation programs, which simultaneously target parent MI and child well-being, yield impacts that are 50% larger in promoting positive child outcomes compared to programs focused solely on addressing parental MI. There is a clear need to provide accessible and scalable solutions that promote positive mental health and developmental outcomes in at-risk children. Digital mental health interventions offer a potential avenue for addressing family needs and barriers to care that are an accessible and low-cost option, and research shows great promise for treating adult depression using these methods. Additional emerging research highlights the efficacy of app-based programs in improving parental MI and parent-child interactions. However, very limited existing app-based or mHealth programs address both parental mental health and parenting skills, which indirectly targets child well-being.

In response to this need, the investigators conducted qualitative research (i.e., focus groups and individual interviews with parents with lived experience) and consulted with a parent advisory board to co-develop a program that simultaneously addressed parental MI and parenting. Results suggested that parents wanted accessible, online services grounded in expert research. Alongside patient-partners and community providers the investigators then developed the BEAM (Building Emotional Awareness and Mental Health) app-based program. The BEAM program is aligned with best practices in mHealth programs including patient-driven priorities, rapid-cycle iterations to facilitate continual improvements, and a commitment to evidenced-based care. Key elements of the original BEAM program include: (1) expert-led educational videos using transdiagnostic therapy and emotion-focused parenting strategies; (2) brief group sessions to consolidate therapeutic content and build social support; (3) a community forum to enhance social connection; and (4) symptom monitoring to track progress. In case of a mental health or parenting-related crisis, clinical coaches also consult via phone. BEAM builds on evidence from the investigative team's knowledge synthesis work suggesting that mHealth therapeutics can address parent MI and while appealing to parents.

The BEAM intervention has consistently demonstrated promising outcomes across various trials to date. The investigative team's latest phase II RCT with mothers of toddlers found that the BEAM program outperformed a services-as-usual (SAU) control condition. Significant improvements in parental MI symptoms including anxiety, anger, and alcohol use were observed. Additionally, BEAM was effective in reducing harsh parenting practices and negative parent-child interactions, with substantial improvements observed for families living in poverty. This trial also showed noteworthy participant engagement with retention rates (84%), comparable to in-person therapy sessions. This phase of research built on and replicated the success of earlier trials with both an open pilot and pilot RCT demonstrating BEAM's efficacy in reducing MI symptoms such as depression, anxiety, anger, sleep issues, and substance use. Qualitative feedback from the initial trials emphasized the positive impact of the BEAM program on mental health and parenting, leading to enhanced quality of life and improved family relationships. Participants also highlighted the value of the social support gained through the online community.

To further address family mental health needs, this trial will test the readiness of the BEAM program for scalability. The current study involves a hybrid effectiveness-implementation trial design to build on previous work. The investigators will use both effectiveness and implementation metrics including short-term follow ups of primary outcomes alongside longer-term follow-ups of mental health and socio-developmental outcomes with linked administrative data. This hybrid design follows the "type 2" model, in which effectiveness and implementation are co-primary aims and can be tracked simultaneously as the trial progresses. This approach is consistent with the investigative team's rapid-cycle program development to date in which BEAM has been tested and adapted in response to patient and provider feedback through each iteration.

This implementation trial aims to maximize BEAM's accessibility, equitability, and effectiveness for future nation-wide implementation. For the current implementation trial, the investigators conducted a full App rebuild to create BEAM Version 2.0 based on participant and Parent Advisory Board feedback. BEAM 2.0 updates include improvements to psychoeducational video content (e.g. high-quality video production, animations, closed captioning), the mobile application user experience (e.g. push notifications, direct messaging, integrated video player that adjusts video quality based on available bandwidth, easy-to-navigate platform), and functionality across mobile device operating systems (iOS, Android). The weekly psychoeducational videos, short symptom tracking surveys, and social support community forum are now housed seamlessly within the BEAM app. Other aspects of the program include individual check ins with trained peer coaches, group drop-in sessions, and a connection to a systems navigator, whose role will be to support participants in accessing community resources.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe symptoms of depression, anxiety, parenting stress, and/or anger (as measured by the PHQ-9, GAD-7, PSI, and PROMIS-Anger). Those who do not have moderate to severe symptoms will meet with a member of the program research team to determine eligibility. This eligibility decision will be based on clinical judgement, ensuring that those with need can participate.
2. Being a parent or primary caregiver of any gender to an 24- to 71-month-old (i.e., 2-5 year old) child.
3. Living in Manitoba.
4. Able to participate in check ins (15 to 60 minutes) via Zoom, phone, direct messaging with a parent peer coach.
5. 18 years or older.
6. Able to understand/read/speak in English.
7. Willing to complete four 45-min questionnaires.
8. At eligibility screening, a question asks if participants have access to an electronic device for viewing videos and participating in Zoom meetings. Participants who do not have access will be asked to contact the research team. The team may be able to accommodate a limited number of participants by providing relevant devices for the duration of the study.
9. Participants have IP addresses within Manitoba, Canada, as determined by IP address in REDCap at time of eligibility screener questionnaire completion. Participants will be required to securely upload a photo that includes both a valid piece of Manitoba government identification and the participant's face (i.e., a 'selfie').

Exclusion Criteria:

1. Living outside of Manitoba.
2. Being a parent or primary caregiver to a child outside of the ages of 24- to 71-months (i.e., 2-5 years).
3. Previously participated in an earlier BEAM trial.
4. Parents who report self-harm that required medical attention within the past six months or a suicide attempt within the past year will be ineligible to participate in BEAM unless the participant is engaged in individual therapy that attends to this acute risk level with one of the following professionals for the duration of the BEAM program: psychiatrist, psychologist, social worker, or psychotherapist. The research team will email all prospective participants who are pending eligibility to schedule a phone call. This call will determine whether it is feasible to connect the participant with an individual therapist to manage specific needs before engaging in the BEAM program, and discuss if the BEAM program is the right fit for the participant's present needs.

Co-parents will be permitted to participate in BEAM regardless of current mental health challenges. Therefore, co-parents are only subject to inclusion criterion (3) and criteria (5-9). Instead of meeting inclusion criteria (2), parenting partners must be a "co-parent (e.g., the child's mom, dad, step-parent) or other primary caregiver (e.g., the child's grandma, cousin, uncle, auntie)" to the corresponding participant's 24- to 71-month-old (i.e., 2-5 year old) child. Co-parents will not receive the same pre-trial screening as parent participants, and thus will not be subject to exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in parent mental health symptom composite. | All measures to be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  The parent mental health composite score will be defined uniquely for each participant using a weighted average of their pre-intervention (T1) mental health profile (i.e., self-report symptoms of depression, anxiety, anger, sleep problems, and parenting stress). Pre-intervention symptoms above established clinical cut-offs will be mean-centred, standardized, and included in the participant's composite mental health symptom score weighted by the symptom's pre-intervention severity. In this way, the primary outcome will track mean change in each participant's most clinically elevated pre-intervention symptoms.
  This composite will use validated measures of depression symptom severity (Patient Health Questionnaire-9), anxiety symptom severity (Generalized Anxiety Disorder-7), anger (PROMIS Anger), sleep disturbances (PROMIS Sleep Disturbance), and parenting stress (Parenting Stress Index - 4th Edition - Short Form). Change in each measure is also a secondary outcome, described below.
Feasibility of the BEAM program. | To be assessed immediately after intervention (T2).
  Feasibility of the BEAM program will be assessed using the mHealth App Usability Questionnaire (MAUQ). The MAUQ is a self-report measure with three subscales that rate ease of use (scores range from 5-35), interface and satisfaction (scores range from 7-49), and usefulness (scores range from 6-42), where high scores indicate better useability.
Acceptability and uptake of the BEAM program. | To be assessed pre-intervention (T1), during intervention, and immediately after intervention (T2).
  Acceptability and uptake of the BEAM program will be assessed in three ways: (1) rates of attrition, (2) qualitative analysis of responses to post-intervention focus group questions that probe barriers and facilitators to program engagement, and (3) program engagement measures from back-end app data (e.g., number of logins, time spent on the app, forum posts, coach engagement, drop-in session engagement, and systems navigator engagement).

SECONDARY OUTCOMES:
Change in parent depressive symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Parent depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a self-report measure of depression symptom severity. Total scores range from 0 to 27, with higher scores indicating more severe depression symptoms.
Change in parent anxiety symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Parent anxiety symptoms will be measured using the Generalized Anxiety Disorder questionnaire (GAD-7). The GAD-7 is a self-report measure of anxiety symptom severity. Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Change in parent anger symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Parent anger symptoms will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anger scale. The PROMIS-Anger is a self-report measure of anger symptoms. Total scores range from 5 to 25, with higher scores indicating more anger symptoms.
Change in parent sleep problems. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Parent sleep problems will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance scale. The PROMIS-Sleep Disturbance is a self-report measure of sleep disturbances. Total scores range from 8 to 40, with higher scores indicating more severe sleep disturbances.
Change in parent alcohol use. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Parent anxiety symptoms will be measured using the Alcohol Use Disorders Identification Test (AUDIT). The AUDIT is a self-report measure of alcohol consumption frequency, drinking behaviors, and frequency of alcohol-related psychological features. Total scores range from 0 to 40, with higher scores indicating more severe alcohol use problems.
Change in parent cannabis use. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Parent anxiety symptoms will be measured using the Cannabis Use Disorders Identification Test-Revised (CUDIT-R). The CUDIT-R is a self-report measure of cannabis consumption frequency, problems, dependence, and cannabis-related psychological features. Total scores range from 0 to 40, with higher scores indicating more severe cannabis use problems.
Change in parenting stress. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Parenting stress will be measured using the Parenting Stress Index - 4th Edition - Short Form (PSI-4-SF). The PSI-4-SF is a self-report measure that captures three sources of stress; from parent stress, from a difficult child, and from parent-child interactions. Total scores range from 36 to 180, with higher scores indicating more parenting stress.
Change in harsh parenting disciplinary practices. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Harsh parenting practices will be measured using 10 items measuring Overreactivity from The Parenting Scale (PS-Overreactivity). The PS-Overreactivity is a self-report measure of parenting behavior and dysfunctional discipline in parents with young children. Total scores range from 10 to 70, with higher scores indicating higher levels of ineffective discipline practices.
Change in child mental health symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Child mental health symptoms will be measured using the Child Behavior Checklist (CBCL). The CBCL is a parent-report measure of emotional and behavioral problems in children. Total scores range from 0 to 198, with higher scores indicating more mental health challenges.
Change in child socioemotional development. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Child socioemotional development will be measured using the Ages and Stages Questionnaires: Socioemotional, Second Edition (ASQ:SE-2). The ASQ:SE-2 is a screening tool that identifies socioemotional challenges across a range of developmental domains. The number of items on the ASQ:SE-2 depend on the age of the child. Higher scores represent more severe socioemotional challenges.
Change in child development. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Child development will be measured using the Ages and Stages Questionnaire, Third Edition (ASQ-3). The ASQ-3 is a parent-report screening tool that measures child developmental progress across domains of communication, motor, problem solving, and personal-social. The number of items on the ASQ:SE-2 depend on the age of the child. Higher scores represent a greater number of met developmental milestones and greater school readiness.

OTHER OUTCOMES:
Change in parenting self-efficacy. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Parenting self-efficacy will be measured using 4 items from the Parenting Stress Index - 4th Edition - Short Form (PSI-4-SF). These 4 items measure parenting self-efficacy. Total scores range from 4 to 20, with higher scores indicating less parenting self-efficacy.
Change in social support. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3), and at 12-month follow-up (T4).
  Social support will be measured using the Social Support Effectiveness Questionnaire (SSEQ). The SSEQ is a self-report measure of partner support effectiveness. Total scores range from 0 to 80, with higher scores indicating greater partner support effectiveness.
Discriminatory experiences. | To be assessed pre-intervention (T1).
  Discrimination will be measured using the Everyday Discrimination Scale (EDS). The EDS is a self-report measure of discriminatory experiences. Total scores range from 0 to 54, with higher scores indicating more discriminatory experiences. This measure may be used as an exploratory mediator or moderator of change.
Adverse childhood experiences. | To be assessed pre-intervention (T1).
  Adverse childhood experiences will be measured using the Adverse Childhood Experiences questionnaire (ACEs). The ACEs is a self-report measure of experiences from childhood that may have been neglectful, abusive, or violent. Total scores range from 0 to 10, with higher scores indicating more adverse childhood experiences. This measure may be used as an exploratory mediator or moderator of change.
Therapeutic alliance. | To be assessed immediately after intervention (T2).
  Therapeutic alliance between peer coaches and participants will be assessed using the Brief Revised Working Alliance Inventory (BR-WAI). The BR-WAI is a 16-item measure assessing bonds, tasks, and goals within the therapeutic relationship. Higher scores indicate stronger alliance. This measure may be used as an exploratory mediator or moderator of change.
Change in administrative measures of family health, education, and social service use. | Administrative data will be drawn from date of childbirth (age 0) to age 8.
  Government records from the Manitoba Population Research Data Repository will assess change in family health, education, and social service use from age 0 to 8. The Families First Home Screening Form assesses perinatal health conditions, perinatal substance use. Mental Health Management Information System assesses parent and child mental illness, mental health service access. Hospital Abstracts Data measures parent and child physical illness, hospitalizations, emergency room visits. Manitoba Immunization Monitoring System assesses vaccination history. Drug Program Information Network measures medication prescribed. Early Developmental Instrument assesses language development, social competence. Enrollment, Marks, and Assessment measures age-appropriate grade, literacy/numeracy in grade 3. Manitoba Education Special Needs assesses if the child has been allotted special needs funding by the province of Manitoba. Vital Statistics Mortality Registry Data measures cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie E Roos, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba - Department of Psychology & Pediatrics, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Summary statistics (e.g., questionnaire subscales, sociodemographics, aggregated forum usage data) paired with non-identifiable participant IDs may be shared on data repositories such as the Open Science Framework.

REFERENCES:
- [Background] Keller PS, Kouros CD, Erath SA, Dahl RE, El-Sheikh M. Longitudinal relations between maternal depressive symptoms and child sleep problems: the role of parasympathetic nervous system reactivity. J Child Psychol Psychiatry. 2014;55(2):172-9. doi: 10.1111/jcpp.12151. Epub 2013 Oct 9. PMID 24117807
- [Background] McGrath JM, Records K, Rice M. Maternal depression and infant temperament characteristics. Infant Behav Dev. 2008 Jan;31(1):71-80. doi: 10.1016/j.infbeh.2007.07.001. Epub 2007 Aug 21. PMID 17714790
- [Background] Skipstein A, Janson H, Kjeldsen A, Nilsen W, Mathiesen KS. Trajectories of maternal symptoms of depression and anxiety over 13 years: the influence of stress, social support, and maternal temperament. BMC Public Health. 2012 Dec 27;12:1120. doi: 10.1186/1471-2458-12-1120. PMID 23270506
- [Background] Mensah FK, Kiernan KE. Parents' mental health and children's cognitive and social development: families in England in the Millennium Cohort Study. Soc Psychiatry Psychiatr Epidemiol. 2010 Nov;45(11):1023-35. doi: 10.1007/s00127-009-0137-y. Epub 2009 Oct 13. PMID 19823757
- [Background] Goodman SH, Rouse MH, Connell AM, Broth MR, Hall CM, Heyward D. Maternal depression and child psychopathology: a meta-analytic review. Clin Child Fam Psychol Rev. 2011 Mar;14(1):1-27. doi: 10.1007/s10567-010-0080-1. PMID 21052833
- [Background] Kingston D, Kehler H, Austin MP, Mughal MK, Wajid A, Vermeyden L, Benzies K, Brown S, Stuart S, Giallo R. Trajectories of maternal depressive symptoms during pregnancy and the first 12 months postpartum and child externalizing and internalizing behavior at three years. PLoS One. 2018 Apr 13;13(4):e0195365. doi: 10.1371/journal.pone.0195365. eCollection 2018. PMID 29652937
- [Background] Azak S, Raeder S. Trajectories of parenting behavior and maternal depression. Infant Behav Dev. 2013 Jun;36(3):391-402. doi: 10.1016/j.infbeh.2013.03.004. Epub 2013 Apr 17. PMID 23603820
- [Background] Vliegen N, Casalin S, Luyten P. The course of postpartum depression: a review of longitudinal studies. Harv Rev Psychiatry. 2014 Jan-Feb;22(1):1-22. doi: 10.1097/HRP.0000000000000013. PMID 24394219
- [Background] Moreno C, Wykes T, Galderisi S, Nordentoft M, Crossley N, Jones N, Cannon M, Correll CU, Byrne L, Carr S, Chen EYH, Gorwood P, Johnson S, Karkkainen H, Krystal JH, Lee J, Lieberman J, Lopez-Jaramillo C, Mannikko M, Phillips MR, Uchida H, Vieta E, Vita A, Arango C. How mental health care should change as a consequence of the COVID-19 pandemic. Lancet Psychiatry. 2020 Sep;7(9):813-824. doi: 10.1016/S2215-0366(20)30307-2. Epub 2020 Jul 16. PMID 32682460
- [Background] Hansen AS, Telleus GK, Mohr-Jensen C, Lauritsen MB. Parent-perceived barriers to accessing services for their child's mental health problems. Child Adolesc Psychiatry Ment Health. 2021 Jan 29;15(1):4. doi: 10.1186/s13034-021-00357-7. PMID 33514400
- [Background] Sztein DM, Koransky CE, Fegan L, Himelhoch S. Efficacy of cognitive behavioural therapy delivered over the Internet for depressive symptoms: A systematic review and meta-analysis. J Telemed Telecare. 2018 Sep;24(8):527-539. doi: 10.1177/1357633X17717402. Epub 2017 Jul 11. PMID 28696153
- [Background] Larkin F, Oostenbroek J, Lee Y, Hayward E, Meins E. Proof of concept of a smartphone app to support delivery of an intervention to facilitate mothers' mind-mindedness. PLoS One. 2019 Aug 22;14(8):e0220948. doi: 10.1371/journal.pone.0220948. eCollection 2019. PMID 31437173
- [Background] Catuara-Solarz S, Skorulski B, Estella-Aguerri I, Avella-Garcia CB, Shepherd S, Stott E, Hemmings NR, Ruiz de Villa A, Schulze L, Dix S. The Efficacy of "Foundations," a Digital Mental Health App to Improve Mental Well-being During COVID-19: Proof-of-Principle Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Jul 1;10(7):e30976. doi: 10.2196/30976. PMID 34978535
- [Background] Roos LE, Kaminski L, Stienwandt S, Hunter S, Giuliano R, Mota N, Katz LY, Zalewski M. The Building Regulation in Dual-Generations Program (BRIDGE): A Mixed-Methods Feasibility Pilot of a Parenting Program for Depressed Mothers of Preschoolers, Matched with Dialectical Behavior Therapy Skills. Child Psychiatry Hum Dev. 2023 Feb;54(1):34-50. doi: 10.1007/s10578-021-01219-1. Epub 2021 Aug 4. PMID 34347227
- [Background] Cameron EE, Simpson KM, Pierce SK, Penner KE, Beyak A, Gomez I, Bowes JM, Reynolds KA, Tomfohr-Madsen LM, Roos LE. Paternal Perinatal Experiences during the COVID-19 Pandemic: A Framework Analysis of the Reddit Forum Predaddit. Int J Environ Res Public Health. 2023 Mar 1;20(5):4408. doi: 10.3390/ijerph20054408. PMID 36901417
- [Background] MacKinnon AL, Silang K, Penner K, Zalewski M, Tomfohr-Madsen L, Roos LE. Promoting Mental Health in Parents of Young Children Using eHealth Interventions: A Systematic Review and Meta-analysis. Clin Child Fam Psychol Rev. 2022 Sep;25(3):413-434. doi: 10.1007/s10567-022-00385-5. Epub 2022 Feb 20. PMID 35184262
- [Background] Barlow DH, Farchione TJ, Bullis JR, Gallagher MW, Murray-Latin H, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Conklin LR, Boswell JF, Ametaj A, Carl JR, Boettcher HT, Cassiello-Robbins C. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders Compared With Diagnosis-Specific Protocols for Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):875-884. doi: 10.1001/jamapsychiatry.2017.2164. PMID 28768327
- [Background] Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Thompson-Hollands J, Carl JR, Gallagher MW, Barlow DH. Unified protocol for transdiagnostic treatment of emotional disorders: a randomized controlled trial. Behav Ther. 2012 Sep;43(3):666-78. doi: 10.1016/j.beth.2012.01.001. Epub 2012 Jan 18. PMID 22697453
- [Background] Spence SH, March S, Donovan CL. Social support as a predictor of treatment adherence and response in an open-access, self-help, internet-delivered cognitive behavior therapy program for child and adolescent anxiety. Internet Interv. 2019 Aug 22;18:100268. doi: 10.1016/j.invent.2019.100268. eCollection 2019 Dec. PMID 31890621
- [Background] Yardley L, Spring BJ, Riper H, Morrison LG, Crane DH, Curtis K, Merchant GC, Naughton F, Blandford A. Understanding and Promoting Effective Engagement With Digital Behavior Change Interventions. Am J Prev Med. 2016 Nov;51(5):833-842. doi: 10.1016/j.amepre.2016.06.015. PMID 27745683
- [Background] Silang KA, Sohal PR, Bright KS, Leason J, Roos L, Lebel C, Giesbrecht GF, Tomfohr-Madsen LM. eHealth Interventions for Treatment and Prevention of Depression, Anxiety, and Insomnia During Pregnancy: Systematic Review and Meta-analysis. JMIR Ment Health. 2022 Feb 21;9(2):e31116. doi: 10.2196/31116. PMID 35188471
- [Background] Swift JK, Greenberg RP. Premature discontinuation in adult psychotherapy: a meta-analysis. J Consult Clin Psychol. 2012 Aug;80(4):547-59. doi: 10.1037/a0028226. Epub 2012 Apr 16. PMID 22506792
- [Background] Xie EB, Freeman M, Penner-Goeke L, Reynolds K, Lebel C, Giesbrecht GF, Rioux C, MacKinnon A, Sauer-Zavala S, Roos LE, Tomfohr-Madsen L. Building Emotional Awareness and Mental Health (BEAM): an open-pilot and feasibility study of a digital mental health and parenting intervention for mothers of infants. Pilot Feasibility Stud. 2023 Feb 18;9(1):27. doi: 10.1186/s40814-023-01245-x. PMID 36800982
- [Background] MacKinnon AL, Simpson KM, Salisbury MR, Bobula J, Penner-Goeke L, Berard L, Rioux C, Giesbrecht GF, Giuliano R, Lebel C, Protudjer JLP, Reynolds K, Sauer-Zavala S, Soderstrom M, Tomfohr-Madsen LM, Roos LE. Building Emotional Awareness and Mental Health (BEAM): A Pilot Randomized Controlled Trial of an App-Based Program for Mothers of Toddlers. Front Psychiatry. 2022 Jun 24;13:880972. doi: 10.3389/fpsyt.2022.880972. eCollection 2022. PMID 35815022
- [Background] Landes SJ, McBain SA, Curran GM. Reprint of: An introduction to effectiveness-implementation hybrid designs. Psychiatry Res. 2020 Jan;283:112630. doi: 10.1016/j.psychres.2019.112630. Epub 2019 Nov 10. PMID 31722790
- [Background] Knapp M, Wong G. Economics and mental health: the current scenario. World Psychiatry. 2020 Feb;19(1):3-14. doi: 10.1002/wps.20692. PMID 31922693
- [Background] McBrien KA, Manns B. Approach to economic evaluation in primary care: review of a useful tool for primary care reform. Can Fam Physician. 2013 Jun;59(6):619-27. PMID 23766042
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Joint Task Force for the Development of Telepsychology Guidelines for Psychologists. Guidelines for the practice of telepsychology. Am Psychol. 2013 Dec;68(9):791-800. doi: 10.1037/a0035001. No abstract available. PMID 24341643
- [Background] Schueller SM, Neary M, Lai J, Epstein DA. Understanding People's Use of and Perspectives on Mood-Tracking Apps: Interview Study. JMIR Ment Health. 2021 Aug 11;8(8):e29368. doi: 10.2196/29368. PMID 34383678
- [Background] Linardon J, Cuijpers P, Carlbring P, Messer M, Fuller-Tyszkiewicz M. The efficacy of app-supported smartphone interventions for mental health problems: a meta-analysis of randomized controlled trials. World Psychiatry. 2019 Oct;18(3):325-336. doi: 10.1002/wps.20673. PMID 31496095
- [Background] Gan DZQ, McGillivray L, Han J, Christensen H, Torok M. Effect of Engagement With Digital Interventions on Mental Health Outcomes: A Systematic Review and Meta-Analysis. Front Digit Health. 2021 Nov 4;3:764079. doi: 10.3389/fdgth.2021.764079. eCollection 2021. PMID 34806079
- [Background] Hanish AE, Lin-Dyken DC, Han JC. PROMIS Sleep Disturbance and Sleep-Related Impairment in Adolescents: Examining Psychometrics Using Self-Report and Actigraphy. Nurs Res. 2017 May/Jun;66(3):246-251. doi: 10.1097/NNR.0000000000000217. PMID 28448375
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Adamson SJ, Kay-Lambkin FJ, Baker AL, Lewin TJ, Thornton L, Kelly BJ, Sellman JD. An improved brief measure of cannabis misuse: the Cannabis Use Disorders Identification Test-Revised (CUDIT-R). Drug Alcohol Depend. 2010 Jul 1;110(1-2):137-43. doi: 10.1016/j.drugalcdep.2010.02.017. Epub 2010 Mar 26. PMID 20347232
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Vaishnavi S, Connor K, Davidson JR. An abbreviated version of the Connor-Davidson Resilience Scale (CD-RISC), the CD-RISC2: psychometric properties and applications in psychopharmacological trials. Psychiatry Res. 2007 Aug 30;152(2-3):293-7. doi: 10.1016/j.psychres.2007.01.006. Epub 2007 Apr 25. PMID 17459488
- [Background] Bjureberg J, Ljotsson B, Tull MT, Hedman E, Sahlin H, Lundh LG, Bjarehed J, DiLillo D, Messman-Moore T, Gumpert CH, Gratz KL. Development and Validation of a Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16. J Psychopathol Behav Assess. 2016 Jun;38(2):284-296. doi: 10.1007/s10862-015-9514-x. Epub 2015 Sep 14. PMID 27239096
- [Background] Orpana HM, Lang JJ, Yurkowski K. Validation of a brief version of the Social Provisions Scale using Canadian national survey data. Health Promot Chronic Dis Prev Can. 2019 Dec;39(12):323-332. doi: 10.24095/hpcdp.39.12.02. PMID 31825785
- [Background] Funk JL, Rogge RD. Testing the ruler with item response theory: increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. J Fam Psychol. 2007 Dec;21(4):572-83. doi: 10.1037/0893-3200.21.4.572. PMID 18179329
- [Background] Williams DR, Yan Yu, Jackson JS, Anderson NB. Racial Differences in Physical and Mental Health: Socio-economic Status, Stress and Discrimination. J Health Psychol. 1997 Jul;2(3):335-51. doi: 10.1177/135910539700200305. PMID 22013026
- [Background] Xie EB, Simpson KM, Reynolds KA, Giuliano RJ, Protudjer JLP, Soderstrom M, Sauer-Zavala S, Giesbrecht GF, Lebel C, Mackinnon AL, Rioux C, Penner-Goeke L, Freeman M, Salisbury MR, Tomfohr-Madsen L, Roos LE. Correction: Building Emotional Awareness and Mental Health (BEAM): study protocol for a phase III randomized controlled trial of the BEAM app-based program for mothers of children 18-36 months. Trials. 2022 Sep 30;23(1):832. doi: 10.1186/s13063-022-06760-5. No abstract available. PMID 36180923
- [Background] Narayan AJ, Rivera LM, Bernstein RE, Harris WW, Lieberman AF. Positive childhood experiences predict less psychopathology and stress in pregnant women with childhood adversity: A pilot study of the benevolent childhood experiences (BCEs) scale. Child Abuse Negl. 2018 Apr;78:19-30. doi: 10.1016/j.chiabu.2017.09.022. Epub 2017 Oct 6. PMID 28992958
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Zhou L, Bao J, Setiawan IMA, Saptono A, Parmanto B. The mHealth App Usability Questionnaire (MAUQ): Development and Validation Study. JMIR Mhealth Uhealth. 2019 Apr 11;7(4):e11500. doi: 10.2196/11500. PMID 30973342
- [Background] Mallinckrodt B, Tekie YT. Item response theory analysis of Working Alliance Inventory, revised response format, and new Brief Alliance Inventory. Psychother Res. 2016 Nov;26(6):694-718. doi: 10.1080/10503307.2015.1061718. Epub 2015 Nov 7. PMID 26549302
- [Background] Smith JD, Stormshak EA, Kavanagh K. Results of a pragmatic effectiveness-implementation hybrid trial of the Family Check-up in community mental health agencies. Adm Policy Ment Health. 2015 May;42(3):265-78. doi: 10.1007/s10488-014-0566-0. PMID 24927926
- [Background] Flight L, Allison A, Dimairo M, Lee E, Mandefield L, Walters SJ. Recommendations for the analysis of individually randomised controlled trials with clustering in one arm - a case of continuous outcomes. BMC Med Res Methodol. 2016 Nov 29;16(1):165. doi: 10.1186/s12874-016-0249-5. PMID 27899073
- [Background] Wall-Wieler E, Roos LL, Nickel NC, Chateau D, Brownell M. Mortality Among Mothers Whose Children Were Taken Into Care by Child Protection Services: A Discordant Sibling Analysis. Am J Epidemiol. 2018 Jun 1;187(6):1182-1188. doi: 10.1093/aje/kwy062. PMID 29617918
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. PLoS Med. 2010 Mar 24;7(3):e1000251. doi: 10.1371/journal.pmed.1000251. PMID 20352064
- [Background] Kwok OM, Underhill AT, Berry JW, Luo W, Elliott TR, Yoon M. Analyzing Longitudinal Data with Multilevel Models: An Example with Individuals Living with Lower Extremity Intra-articular Fractures. Rehabil Psychol. 2008 Aug;53(3):370-386. doi: 10.1037/a0012765. PMID 19649151
- [Background] Archibald M, Wiebe S, Rieger K, Linton J, Woodgate R. Protocol for a systematic review of living labs in healthcare. BMJ Open. 2021 Feb 5;11(2):e039246. doi: 10.1136/bmjopen-2020-039246. PMID 33550226
- [Background] Archibald MM, Wittmeier K, Gale M, Ricci F, Russell K, Woodgate RL. Living labs for patient engagement and knowledge exchange: an exploratory sequential mixed methods study to develop a living lab in paediatric rehabilitation. BMJ Open. 2021 May 4;11(5):e041530. doi: 10.1136/bmjopen-2020-041530. PMID 33947723
- [Background] Kim J, Kim YL, Jang H, Cho M, Lee M, Kim J, Lee H. Living labs for health: an integrative literature review. Eur J Public Health. 2020 Feb 1;30(1):55-63. doi: 10.1093/eurpub/ckz105. PMID 31169898
- [Background] Farmer AY, Lee SK. The effects of parenting stress, perceived mastery, and maternal depression on parent-child interaction. Journal of Social Service Research. 2011; 37(5): 516-525.
- [Background] Lipscomb ST, Hatfield B, Lewis H, Goka-Dubose E, Fisher PA. Strengthening children's roots of resilience: Trauma-responsive early learning. Children and Youth Services Review. 2019; 107: 104510.
- [Background] Lambert MJ, Harmon KL. The merits of implementing routine outcome monitoring in clinical practice. Clinical Psychology: Science and Practice. 2018; 25(4): e12268.
- [Background] Arnold DS, O'Leary SG, Wolff LS, Acker MM. The Parenting Scale: A measure of dysfunctional parenting in discipline situations. Psychological Assessment. 1993; 5(2): 137-144.
- [Background] Rini C, Schetter CD, Hobel CJ, Glynn LM, Sandman CA. Effective social support: Antecedents and consequences of partner support during pregnancy. Personal Relationships. 2006; 13(2): 207-229.
- [Background] Patton MQ. Qualitative research & evaluation methods. 3rd ed. Thousand Oaks: Sage; 2010.
- [Background] Enders CK. Applied missing data analysis. 2nd ed. The Guilford Press; 2022.
- [Background] Pierce S, de Castro Lima HL, Jain B, Reynolds KA, Tomfohr-Madsen LM, Roos LE. A unique role for social connextion in the COVID-19 pandemic; a qualitative analysis of parenting forums. Center for Open Science. Preprint posted online February 5, 2022.
- [Background] Flannery J, Penner-Goeke L, Xie EB, Prince D, Simpson KM, Callaghan B, Tomfohr-Madsen L, Roos LE. Digital parent training RCT meta-analysis and semantic review. PsyArXiv. Preprint posted online January 15, 2021. osf.io/cpd9b
- [Background] Roos LE, MacKinnon AL, Xie EB, Simpson KM, Rioux C, Reynolds KA, et al. Treating maternal mental health problems with an app-based program: A randomized control trial of BEAM, for mothers of young children. Submitted 2023.
- [Background] Abidin RR. Parenting stress index. 4th Edition. Psychological Assessment Resources, Inc.; 2012.
- [Background] Achenbach TM, Rescorla L. Manual for the ASEBA school-age forms & profiles: an integrated system of multi-informant assessment. Burlington, VT: ASEBA; 2001.
- [Background] Squires J, Bricker DD, Twombly E. Ages & stages questionnaires, social-emotional (ASQ:SE-2TM)): a parent-completed child monitoring system for social-emotional behaviors. Second edition. Baltimore, Maryland: Brookes Publishing; 2015.
- [Derived] Simpson KM, McHardy RJW, Zhou JG, Levasseur-Puhach S, Cote CM, Braun M, Clement F, MacKinnon AL, Nickel N, Afifi TO, Giesbrecht GF, Giuliano R, Katz LY, Kelly LE, Klassen TP, Lebel C, Mushquash A, Reynolds K, Decaire E, Mughal W, Chartrand F, Kloss O, Hensel JM, Bolton JM, Unger JAM, Archibald M, Fisher P, Pharazyn A, Tomfohr-Madsen L, Roos LE. Building Emotional Awareness and Mental Health (BEAM): study protocol for a hybrid implementation-effectiveness trial of the BEAM app-based program for parents with clinical mental health problems. BMC Psychiatry. 2025 Jun 2;25(1):567. doi: 10.1186/s12888-025-06964-4. PMID 40457257
- See also: Statistics Canada. Leading causes of death, total population, by age group [Internet]. Government of Canada; [accessed 2024 Jan 14] — https://www150.statcan.gc.ca/t1/tbl1/en/tv.action?pid=1310039401
- See also: Health Canada. Canadian Community Health Survey, Cycle 2.2, Nutrition (2004): Income-related household food security in Canada. [Internet]. 2007 — https://www.canada.ca/content/dam/hc-sc/migration/hc-sc/fn-an/alt_formats/hpfb-dgpsa/pdf/surveill/income_food_sec-sec_alim-eng.pdf
- See also: Statistics Canada. Canadian housing survey, 2022. [Internet]. 2022 — https://www23.statcan.gc.ca/imdb/p3Instr.pl?Function=assembleInstr&lang=en&Item_Id=1479765